CLINICAL TRIAL: NCT04753268
Title: Preliminary Examination of a Mobile Behavior Change Program for Weight Loss in Breast Cancer Survivors
Brief Title: Mobile Behavior Change Program for Weight Loss in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noom Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00048814
Record Dates: First submitted 2021-01-29; First posted 2021-02-15 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Weight Loss; Behavior, Health
MeSH Terms: conditions — Weight Loss; Health Behavior

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm pilot study evaluating preliminary efficacy and acceptability of a Noom breast cancer survivor weight loss program.
  The intervention consists of a curriculum, provided through daily articles that users are encouraged to read; logging features for weight, meals, and physical activity; in-app groups; and a virtual coach, who will communicate with participants via in-app messaging. During the first week of the study, participants will be introduced to the program, the Noom app, and their coach.
  Coaches will use a secure dashboard to monitor patient progress, which is used to increase engagement and motivation. Participants are encouraged to log their weight, physical activity, and meals daily.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group: Noom Healthy Weight Program (Experimental): The intervention consists of a curriculum, provided through daily articles that users are encouraged to read; logging features for weight, meals, and physical activity; in-app groups; and a virtual coach, who will communicate with participants via in-app messaging.
  Interventions: Behavioral: Noom Healthy Weight Program

INTERVENTIONS:
Behavioral: Noom Healthy Weight Program — The intervention consists of a curriculum, provided through daily articles that users are encouraged to read; logging features for weight, meals, and physical activity; in-app groups; and a virtual coach, who will communicate with participants via in-app messaging. During the first week of the study, participants will be introduced to the program, the Noom app, and their coach.
  Coaches will use a secure dashboard to monitor patient progress, which is used to increase engagement and motivation. Participants are encouraged to log their weight, physical activity, and meals daily.

SUMMARY:
The purpose of this study is to evaluate the preliminary efficacy of a Noom Breast Cancer Weight Loss Program on weight loss outcomes, quality of life, and physical activity. Also, to qualitatively determine acceptability of this novel program among breast cancer survivors with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent
* 18 years and older
* Overweight or obesity (BMI ≥ 27.5)
* Not 6 months postpartum
* Not planning to become pregnant in the next 7 months
* Have a smartphone that is compatible with Noom's mobile app
* Breast cancer survivor with stage I, II, or III
* Completed active treatment (e.g, surgery, chemo, radiation, etc.) > 6 months ago

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent
* Currently pregnant or < 6 months postpartum
* Plans to become pregnant within the next 7 months
* Stage IV, metastatic cancer or DCIS
* Currently taking insulin
* Uncontrolled hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female survivors of breast cancer
Enrollment: 30 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Weight | baseline to 6 months
  Self-reported weight
Program engagement | weeks 1-26
  Engagement with the Noom program; measured as
  1. Number of App opens
  2. Messages to coach
  3. Number of Steps
  4. Logged food
  5. Logged exercise
  6. Group messages and likes
  7. Articles read
Program retention | weeks 1-26
  i.e. % = (total participants - number of drop out) / Total number of participants) * 100%
Program satisfaction | week 1 - 26 week
  Satisfaction assessed via an in-house survey

CONTACTS AND LOCATIONS:
Locations (1):
- Noom, Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen S, Salehi E, White C, Chen Y, Iyengar NM. Evaluation of a mobile behavior change program for weight loss in breast cancer survivors. NPJ Breast Cancer. 2024 Jun 29;10(1):53. doi: 10.1038/s41523-024-00659-x. PMID 38951532